CLINICAL TRIAL: NCT04251325
Title: Socio-demographic Characteristics of Basic Life Support Course Participants
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Other Study IDs: Socio-demographic BLS
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: BLS; Recruitment

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Basic Life Support Course Participants: The study population includes all Danish citizens who attended a BLS training course certificate from 2016-2018 above the age of 15.
  Interventions: Other: Basic Life Support Courses
- Background population: The entire danish population above 15 years whom have not attended a BLS training course certificate from 2016-2018.

INTERVENTIONS:
Other: Basic Life Support Courses — 4 hours basic life support courses for laypersons
  Groups: Basic Life Support Course Participants

SUMMARY:
Aim The aim of the study is to characterize the typical basic life support (BLS) course participant. The characterization include age, sex, education, ethnicity, income, health care data and cohabitation. All data will be compared with that of the general population. Hereby the study wish identify potential focus areas for recruitment of willing and able bystanders to increase survival. Furthermore, this study will provide a foundation for evaluation of current initiatives.

Significance In Denmark, several population-based campaigns have been initiated to increase the amount of able and willing laypersons to assist at out-of-hospital cardiac arrest (OHCA). The main focus has been on increasing the quantity of laypersons attending BLS courses. Even measures of changing legislation mandating course participation have been passed and implemented. Estimates state that approximately 3-4.5% of the entire Danish population participates in BLS courses annually. Consequently, a substantial amount of resources has been spent on educating and certifying laypersons in BLS on a population level. In this study, the characteristics of these BLS course participants will be described. This will provide the basis for evaluation of already implemented interventions. Additionally, this study will be able to support course distributors, foundations and national councils in making strategies for further recruitment based on evidence. The present study will assist in pinpointing society groups with a theoretical bystander potential, but low level of BLS education. This can guide future efforts in trying to improve bystander initiated cardiopulmonary resuscitation (CPR) and survival from OHCA.

Methods The study population includes all Danish citizens who attended a BLS training course certificate from 2016-2018 above the age of 15. This cut off is based on the earliest mandatory BLS training in primary school. Using Personal Identifications Numbers (PIN) of BLS course participant from January 1st, 2016 to December 31st, 2018, data will be extracted and delivered anonymously, including information on age, sex, income, education, ethnicity and cohabitation, from the Statistics Denmark. The relative risk of BLS course attendance stratified by education and income level, cohabitation status, age of youngest child, urbanization level, sex and ethnicity of the Danish BLS course participants compared to the general population will be presented. Prevalence of BLS courses participants by age and sex will be analyzed and graphically display and prevalence of BLS course participants by income and age will be calculated by regression models. A layperson focus group interview consisting of BLS course participants will be conducted to explore the attending courses participants views of the project and to revise accordingly.

Anonymity is secured through a data processing agreement between the Danish First Aid Council and Statistics Denmark, facilitated by the Copenhagen Emergency Medical Services. An application will be formulated to the Danish Data protection agency regarding storage of data.

Expected outcome A characterization of the typical BLS course participants in Denmark with median age, sex, cohabitation, income and education. The association between sociodemographic characteristics of BLS course participants and relevant prevalence's by the entire population will be presented.

DETAILED DESCRIPTION:
Background Bystander initiated basic life support (BLS) play an increasingly important role in the efforts and strategies to improve survival from out-of-hospital cardiac arrest (OHCA). Denmark is known internationally for our ability to investigate OHCA on a population scale and for the high number of laypersons educated in BLS. Denmark has approximately 5400 OHCA each year.

There has been a significant increase in survival after OHCA in Denmark the last two decades. Since 2001, the 30-day survival rate has increased fourfold from approximately 4% in 2001 to 16% in 2018. This increase has been linked to a significant rise in bystander-initiated CPR prior to the arrival of emergency medical services (EMS).

The Global Resuscitation Alliance emphasizes the need to educate laypersons in BLS and of the ten steps to improve survival from OHCA, four steps involve BLS and the community. It is stated by the Global Resuscitation Alliance that "a population universally trained in CPR has the potential to double survival rates" . Bystander-initiated CPR rate has increased from 20% in 2001 to 77% in 2018. In the same period as Denmark have witnessed a fourfold increase in bystander-initiated CPR and approximately threefold increase in the number of basic life support courses have been seen.

The rise number of basic life support courses in is largely due to several central initiatives. To increase bystander CPR rates in Denmark, CPR courses have been made mandatory in all primary schools since January 2005 and when taking driver's license since October 2006. Further, several large scale national campaigns, like TrygFondens Heartrunners, have been initiated to increase bystander CPR rates and the use of automatic external defibrillators (AED) for laypeople. An examination of TrygFondens First Responders project Heartrunners showed that up to 98% of the first responders had participated in BLS course and a majority (70%) within the last two years. Hence, the soon to be national, first responder project TrygFondens Heartrunners is recruiting largely among citizens whom have participated in BLS courses within the last two years.

Further, in an upcoming study of a representative part of the entire population, 4 out of 5 respondents answered that they had participated in some kind of BLS course in their lifetime. Unverified numbers assert that approximately 250.000-300.000 citizens attend certified BLS courses annually. This entails, that approximately 3-4,5% of the entire Danish population attain a certificate annually. However, the measure of annual BLS course participants in Denmark is, for now, only an assumption. When engaging 3-4.5% of the entire Danish population annually, it is reasonable to evaluate the effort. Little is known about the profile of this large proportion of Danish citizens. Obvious questions to be asked are; "Can the numbers be verified?", "Are the targeted groups of potential bystanders reached?" and "To recruit and maintain able and willing bystanders, whom should campaigns address?"

Most courses (>97%) are provided by one of the organizations of the Danish First Aid Council or the danish Heart Foundation. Only a minor proportion of approximately 2.500-4.000 are provided by the Danish/European resuscitation council. All recognized providers intend to follow the standards of the ERC guidelines. Since 2016 the Danish First Aid Council, who conduct most courses, have registered all certificates electronically with Personal Identification Number (PIN) of participants, type of course and date of passed course for each of the approximately 250.000-300.000 participants annually. The courses include 4 hours training in BLS including CPR and AED use. The Danish Heart Foundation have created a voluntary based BLS introduction course of 30 minutes length including CPR and AED use.

To maintain the high number potential bystanders based on able and willing laypersons to act at OHCA, it is essential to not only retain the active BLS educated able bystanders, but also to continuously recruit new potential able bystanders.

Recruitment efficacy is optimized by targeting those segments of the population with the largest available resource and by focusing on those who are the most likely to respond positively. The willingness to provide BLS by layperson and attending a course has many similarities with the willingness to donate blood. Therefore, it is reasonable to look at initiatives involved in maintaining and increasing recruitment of blood donors on a national level. In a study from 2017 Burgdorf et al. examined the Danish blood donors and assume that potential donors would be similar those who already have donated with respect to age, sex and sociodemographic characteristics. Similarly, it is rational to attain more detailed knowledge of who attend BLS courses to increase and maintain recruitment for current at future BLS educational interventions.

Aim:

1. To characterize the typical BLS course participants. The characterization includes: age, sex, income, education, ethnicity, health care data and cohabitation in comparison with the general population
2. To identify recruitment potentials in the general public for BLS educational interventions to increase survival
3. To provide basis information to be used when designing strategies for recruitment to population-based BLS educational interventions to increase survival

Relevance This study will provide knowledge that can help optimization of public efforts to increase the willingness to help in all emergency situations and specifically increase the knowledge of those willing to aid as bystander for OHCA. By extension this will increase survival. This can result in optimization of future campaigns to improve survival and evaluation of current national population-based interventions.

Methods The study is a registry-based follow-up study. The study population comprised all Danish citizens above the age of 15 in 2018. This cut of is based on earliest mandatory BLS training in school and will have no upper age limit. The methodical approach is in large guided by similar studies examining recruitment potential and characteristics of a population-based effort to increase willingness of laypersons donating blood.

Since 1968 all Danish citizens have been identifiable through a 10-digit Personal Identification Number (PIN). Through Statistics Denmark it is possible to attain sociodemographic data from PIN numbers. When the investigated population is sufficiently large, the data output will be considered anonymously encrypted by the Statistics Denmark.

Statistical analysis data storage and anonymization With the PIN numbers of all BLS course participants, the current study wish to extracted information on sex; year of birth; ethnicity (born in Denmark by at least one ethnically Danish parent, born in Denmark by non-Danish parents, born in a Western country other than Denmark, or born in a non-Western country); parental birth place; cohabitation status (living with parents, living alone, living with a person of opposite gender, living with a person of same gender, living in a multi-household which is a household with three or more unrelated adults); age of youngest child in the household (0, 1-2, 3-5, 6-8, 9-11 or 12+ years old, or no children); and level of urbanization (<25, 25-350, >350-1000, >1000-2000, >2000 persons per square kilometer); education (primary and lower secondary education, high school, technical and vocational education and training, higher short/middle length education, higher long term education), and income (deciles relative to gender and birth year) and potentially health care data (number of hospitalizations and parameters related to general health) as done in previous study on blood donors. For all the above-mentioned parameters reference values for the background population is extracted as reference for direct statistical comparison. To estimate relative risk (RR) or odds ratio (OR) of attending a BLS course for demographic/sociodemographic variables, binary regression models with log-link or multiple logistic regression will be conducted. Maximum likelihood estimate of RR and 95% confidence intervals will be calculated in a joint model. Data are presented with prevalence of BLS course certificate with mutually adjusted RR or OR and 95% confidence intervals. The relative risk for each subgroup is compared to the reference group (RR = 1.00). To show the prevalence as a smooth function of age, this study will identified the number of BLS course certificates and number of potential able bystanders at each age in days or months. If needed the prevalence will smoothed using the loess algorithm.

Data management and statistical analyses will be performed using R-statics™ (The R Foundation for Statistical Computing, Austria). All data will be stored anonymously on secured folder within the regional central IT system. A formal application to Danish data Protection Agency regarding usage, transformation and storage of certificate data will be formulated.

Ethics Because this is a Registry-based study no ethical approval is required. However, the the regional committee for ethical approval have been contacted will register this study with a unique registration number for approval.

ELIGIBILITY:
Inclusion Criteria:

All danish citizens, with a verified personal identification number, whom participated in a certified basic life support course between 2016 and 2019.

Exclusion Criteria:

Basic life support course participants with in-complete/faulty registered personal identification number.

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All danish citizens whom participated in a certified basic life support course between 2016 and 2019.
Sampling Method: Non-Probability Sample
Enrollment: 900000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Sex | 2016-2018
  Male, female
Age | 2016-2018
  In either month or days (to enable smooth curves)
Ethnicity | 2016-2018
  born in Denmark by at least one ethnically Danish parent, born in Denmark by non-Danish parents, born in a Western country other than Denmark, or born in a non-Western country)
Parental birth place | 2016-2018
  Danish region
Cohabitation status | 2016-2018
  Living with parents, living alone, living with a person of opposite gender, living with a person of same gender, living in a multi-household which is a household with three or more unrelated adults
Age of youngest child in the household | 2016-2018
  0, 1-2, 3-5, 6-8, 9-11 or 12+ years old, or no children
Level of urbanization | 2016-2018
  <25, 25-350, >350-1000, >1000-2000, >2000 persons per square kilometer
Education | 2016-2018
  Primary and lower secondary education, high school, technical and vocational education and training, higher short/middle length education, higher long term education
Income | 2016-2018
  Deciles relative to gender and birth year

OTHER OUTCOMES:
Health care data | 2016-2018
  number of hospitalizations and parameters related to general health

CONTACTS AND LOCATIONS:
Overall Officials: Freddy K Lippert, MD,Ass.Prof, Study Chair — Copenhagen Emergency Medical Services
Locations (1):
- Copenhagen Emergency Medical Services, Copenhagen, Denmark

REFERENCES:
- [Background] Eisenberg M, et al. Acting on the Call. 2019 [ONLINE] Available at: http://www.globalresuscitationalliance.org/wp-content/pdf/acting_on_the_call.pdf
- [Background] Eisenberg M, et al. A call to establish a global resuscitation alliance. 2018 [ONLINE] Available at: https://foundation915.files.wordpress.com/2016/07/a-call-to-establish-a-global-resuscitation-alliance-2016.pdf [Accessed November 18 2019].
- [Background] Dansk Hjertestopsregister [Internet/in Danish]. [cited 2019 Nov 06]; Available from: http://hjertestopregister.dk/wp-content/uploads/2019/11/Dansk-Hjertestopregister-2018.pdf
- [Background] Wissenberg M, Lippert FK, Folke F, Weeke P, Hansen CM, Christensen EF, Jans H, Hansen PA, Lang-Jensen T, Olesen JB, Lindhardsen J, Fosbol EL, Nielsen SL, Gislason GH, Kober L, Torp-Pedersen C. Association of national initiatives to improve cardiac arrest management with rates of bystander intervention and patient survival after out-of-hospital cardiac arrest. JAMA. 2013 Oct 2;310(13):1377-84. doi: 10.1001/jama.2013.278483. PMID 24084923
- [Background] Hansen SM, Hansen CM, Folke F, Rajan S, Kragholm K, Ejlskov L, Gislason G, Kober L, Gerds TA, Hjortshoj S, Lippert F, Torp-Pedersen C, Wissenberg M. Bystander Defibrillation for Out-of-Hospital Cardiac Arrest in Public vs Residential Locations. JAMA Cardiol. 2017 May 1;2(5):507-514. doi: 10.1001/jamacardio.2017.0008. PMID 28297003
- [Background] Kragholm K, Wissenberg M, Mortensen RN, Hansen SM, Malta Hansen C, Thorsteinsson K, Rajan S, Lippert F, Folke F, Gislason G, Kober L, Fonager K, Jensen SE, Gerds TA, Torp-Pedersen C, Rasmussen BS. Bystander Efforts and 1-Year Outcomes in Out-of-Hospital Cardiac Arrest. N Engl J Med. 2017 May 4;376(18):1737-1747. doi: 10.1056/NEJMoa1601891. PMID 28467879
- [Background] Hansen CM, Lippert FK, Wissenberg M, Weeke P, Zinckernagel L, Ruwald MH, Karlsson L, Gislason GH, Nielsen SL, Kober L, Torp-Pedersen C, Folke F. Temporal trends in coverage of historical cardiac arrests using a volunteer-based network of automated external defibrillators accessible to laypersons and emergency dispatch centers. Circulation. 2014 Nov 18;130(21):1859-67. doi: 10.1161/CIRCULATIONAHA.114.008850. Epub 2014 Oct 1. PMID 25274002
- [Background] Malta Hansen C, Zinckernagel L, Ersboll AK, Tjornhoj-Thomsen T, Wissenberg M, Lippert FK, Weeke P, Gislason GH, Kober L, Torp-Pedersen C, Folke F. Cardiopulmonary Resuscitation Training in Schools Following 8 Years of Mandating Legislation in Denmark: A Nationwide Survey. J Am Heart Assoc. 2017 Mar 14;6(3):e004128. doi: 10.1161/JAHA.116.004128. PMID 28292745
- [Background] Copenhagen Emergency Medical Services, research presentation [Internet/in Danish]. [cited 2019 Nov 30]; Available from: https://docplayer.dk/159358374-Trygfondens-hjerteloeber-projekt-region-syd-vejle-12-august-2019.html
- [Background] TrygFonden [Internet/in Danish]. [cited 2019 Nov 06]; Available from: https://genoplivning.dk/nyt-studie-4-5-danskere-har-vaeret-paa-foerstehjaelpskursus/
- [Background] Perkins GD, Handley AJ, Koster RW, Castren M, Smyth MA, Olasveengen T, Monsieurs KG, Raffay V, Grasner JT, Wenzel V, Ristagno G, Soar J; Adult basic life support and automated external defibrillation section Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 2. Adult basic life support and automated external defibrillation. Resuscitation. 2015 Oct;95:81-99. doi: 10.1016/j.resuscitation.2015.07.015. Epub 2015 Oct 15. No abstract available. PMID 26477420
- [Background] Burgdorf KS, Simonsen J, Sundby A, Rostgaard K, Pedersen OB, Sorensen E, Nielsen KR, Bruun MT, Frisch M, Edgren G, Erikstrup C, Hjalgrim H, Ullum H. Socio-demographic characteristics of Danish blood donors. PLoS One. 2017 Feb 9;12(2):e0169112. doi: 10.1371/journal.pone.0169112. eCollection 2017. PMID 28182624
- [Background] Ou Y, Yau KK, Poon CM, Hui YV, Lee SS, Lee CK. Donation frequency and its association with demographic characteristics--a 1-year observational study. Transfus Med. 2015 Dec;25(6):366-73. doi: 10.1111/tme.12267. Epub 2016 Jan 5. PMID 26729059
- [Background] Ritter S, Willand L, Reinhard B, Offergeld R, Hamouda O. [Demography and donation frequencies of blood and plasma donor populations in Germany]. Bundesgesundheitsblatt Gesundheitsforschung Gesundheitsschutz. 2008 Aug;51(8):915-25. doi: 10.1007/s00103-008-0613-7. German. PMID 18787870
- [Background] Lattimore S, Wickenden C, Brailsford SR. Blood donors in England and North Wales: demography and patterns of donation. Transfusion. 2015 Jan;55(1):91-9. doi: 10.1111/trf.12835. Epub 2014 Sep 1. PMID 25178387
- [Background] Schmidt M, Schmidt SAJ, Adelborg K, Sundboll J, Laugesen K, Ehrenstein V, Sorensen HT. The Danish health care system and epidemiological research: from health care contacts to database records. Clin Epidemiol. 2019 Jul 12;11:563-591. doi: 10.2147/CLEP.S179083. eCollection 2019. PMID 31372058
- [Background] Cleveland WS. Devlin SJ, and Grosse E. (1988).